CLINICAL TRIAL: NCT01633853
Title: Study of Vitamin D2 Virus 1,25(OH)2-Vitamin D3 in the Treatment of Chronic Kidney Disease Mineral and Bone Disease
Brief Title: Efficacy of Vitamin D2 to Treat Chronic Kidney Disease Mineral and Bone Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dongliang Zhang, MD (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor-Investigator, Dongliang Zhang, MD, Associate Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-078; Z121107001012138 (Other Grant/Funding Number: Beijing Municipal Science and Technology Commission); 2011-2002-02 (Other Grant/Funding Number: The capital health research and development of special)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Vitamin D Deficiency
Keywords: chronic kidney disease mineral and bone disorder; vitamin D2; parathyroid hormone
MeSH Terms: conditions — Vitamin D Deficiency; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Ergocalciferols; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D2 Treatment (Experimental): Patients will be treated by vitamin D2. Oral Vit D2 1.25mg(50,000 unit) once weekly as a start and maintain 1.25mg(50,000 unit) once monthly according to the blood 25(OH)vitamin D level.
  Interventions: Drug: Vitamin D2
- 1,25(OH)2 Vitamin D3 (Active Comparator): Patients will be treated by 1,25(OH)2 Vitamin D3. Oral 1,25(OH)2 Vitamin D3(Rocaltrol) by 0.25 microgram once daily at start and regulate the dose according to the changes of blood levels of 25(OH)Vit D, calcium, phosphorus, and intact parathyroid hormone.
  Interventions: Drug: 1,25(OH)2 Vit D3

INTERVENTIONS:
Drug: Vitamin D2 — Treatment with Vit D2.
  Other Names: Vitamin D2 soft capsules
  Arms: Vitamin D2 Treatment
Drug: 1,25(OH)2 Vit D3 — Treatment with 1,25(OH)2 Vitamin D3(Rocaltrol).
  Other Names: Rocaltrol
  Arms: 1,25(OH)2 Vitamin D3

SUMMARY:
It is hypothesised that the efficacy and safety of Vitamin D2 soft capsule to treat the Chronic Kidney Disease Mineral and Bone Disease (CKD-MBD) are equal to 1,25(OH)2 Vitamin D3 (Rocaltrol) in the patients with CKD stage 3-5.

DETAILED DESCRIPTION:
This study will enroll chronic kidney disease patients, stage 3 to 5, who have chronic kidney disease mineral and bone disease (CKD-MBD)as defined by Kidney Disease Improvement Global Outcome (KDIGO) Guidelines. Patients in one center will be randomized to receive oral Vitamin D2 soft capsule or Rocaltrol. A total of 200 patients will be enrolled, 100 in the Vitamin D2 group and 100 in the 1,25(OH)2 Vitamin D3 group. Outcomes will be assessed as proportion of patients achieving target blood levels on calcium, phosphorus, parathyroid hormone, and 25 hydroxyvitamin D. Other outcomes will also be assessed, which include secondary hyperparathyroidism (sHPT), vascular calcification, and cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18-75 years.
* Patients with chronic kidney disease stage 3 to 5, and concurrent chronic kidney disease mineral and bone disorder.

Exclusion Criteria:

* Renal artery stenosis, inherent renal malformation, solitary kidney, or malignancy in urinary system.
* New fracture in last 3 months.
* Active system immunity diseases.
* History of liver failure
* History of intestinal malabsorption or chronic diarrhea
* Treatment with phenobarbital, phenytoin, rifampicin, sucralfate, steroids, digoxin, or other medications that could affect vitamin D metabolism
* Primary hyperparathyroidism
* Treatment with cinacalcet or other calcimimetic within the past 6 months
* Anticipated dialysis within 6 months after randomization
* Have an unstable medical condition, defined as having been hospitalized within 30 days before screening, the expectation of recurrent hospital admissions or life expectancy of less than 6 months in the judgment of the investigator
* Subject is currently enrolled in, or fewer than 30 days have passed since subject has completed another investigational device or drug study(s); or subject is receiving another investigational agent(s).
* Current treatment with vitamin D 50,000 IU
* Using glucocorticoid or immunosuppressive agents.
* Acute renal dysfunction.
* The expected live time is less than 2 years.
* Pregnant or lactating woman.
* Suffered from acute myocardial infraction, acute congestive heart failure, or stroke in last 6 months.
* Patients whose concurrent illnesses, disability, or geographical residence would hamper attendance at required study visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dongliang Zhang, Doctor, Principal Investigator — Nephrology Department of Beijing Friendship Hospital
Locations (1):
- Beijing Friedship Hospital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D2: Patients will be treated by vitamin D2. Oral Vit D2 1.25mg(50,000 unit) once weekly as a start and maintain 1.25mg(50,000 unit) once monthly according to the blood 25(OH)vitamin D level.
  Vitamin D2: Treatment with Vit D2.
Period: Overall Study
Arm/Group | Vitamin D2 | 1,25(OH)2 Vitamin D3
Started | 104 | 100
Completed | 104 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D2 | 1,25(OH)2 Vitamin D3 | Total
Number analyzed (Participants) | 104 | 100 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.35 (5.64) | 56.27 (5.94) | 56.89 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 74 | 66 | 140
Region of Enrollment [Number; unit: participants]
  China | 104 | 100 | 204
Ca-baseline [Mean (Standard Deviation); unit: mmol/L] | 2.29 (0.14) | 2.31 (0.11) | 2.30 (0.12)
P-baseline [Mean (Standard Deviation); unit: mmol/L] | 1.15 (0.24) | 1.14 (0.21) | 1.14 (0.22)
iPTH-baseline [Mean (Standard Deviation); unit: ng/ml] | 109.7 (127.8) | 89.5 (75.0) | 98.2 (100.1)
25(OH)Vit D [Mean (Standard Deviation); unit: ng/ml] | 15.14 (7.46) | 14.90 (6.15) | 15.02 (6.83)

OUTCOME MEASURES:

1. Primary Outcome: The Blood Levels of Calcium at the 24th Month of Following up.
Description: The blood levels of calcium at the 24th month of following up will be detected.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D2 | 1,25(OH)2 Vitamin D3
Number analyzed (Participants) | 104 | 100
mmol/L | 2.31 (0.14) | 2.33 (0.14)
Statistical Analysis 1: Comparison: Vitamin D2; The blood levels of calcium at the 24th month of following up were compared to the levels of the baseline both in group Vitamin D2; Test type: Superiority or Other; p = 0.117, t-test, 2 sided
Statistical Analysis 2: Comparison: 1,25(OH)2 Vitamin D3; The blood levels of calcium at the 24th month of following up were compared to the levels of the baseline in group 1,25(OH)2 Vitamin D3; Test type: Superiority or Other; p = 0.309, t-test, 2 sided
Statistical Analysis 3: Comparison: Vitamin D2 vs 1,25(OH)2 Vitamin D3; The levels of blood calcium at the 24th month of following up were compared between two groups; Test type: Superiority or Other; p = 0.554, t-test, 2 sided — t=-0.593

2. Secondary Outcome: The Blood 25(OH)Vitamin D Level.
Description: The levels of blood 25(OH)Vitamin D at the 24th month of following up.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vitamin D2 | 1,25(OH)2 Vitamin D3
Number analyzed (Participants) | 104 | 100
ng/ml | 37.31 (10.49) | 18.07 (7.55)
Statistical Analysis 1: Comparison: Vitamin D2 vs 1,25(OH)2 Vitamin D3; The levels of blood 25(OH)Vitamin D were compared between the 24th month and the baseline in group Vitamin D2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1,25(OH)2 Vitamin D3; The levels of blood 25(OH)Vitamin D were compared between the 24th month and the baseline in group 1,25(OH)2 Vitamin D3; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Vitamin D2 vs 1,25(OH)2 Vitamin D3; The levels of blood 25(OH) Vitamin D at the 24th month of following up were compared between two groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P<0.001, t=-14.982

3. Secondary Outcome: The Incidence Rate of Secondary Hyperparathyroidism.
Description: Patients with the blood iPTH level higher than 300 pg/ml will be regard as sHPT. The incidence of sHPT during following up were recorded and compared between two groups.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Vitamin D2 Treatment | 1,25(OH)2 Vitamin D3
Number analyzed (Participants) | 104 | 100
participants | 14 | 15
Statistical Analysis 1: Comparison: Vitamin D2 Treatment vs 1,25(OH)2 Vitamin D3; Test type: Superiority or Other; p = 0.753, Chi-squared — Chi-square value=0.099

4. Primary Outcome: The Blood Levels of Phosphorus at the 24th Month of Following up.
Description: The blood levels of phosphorus at the 24th month of following up will be detected.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D2 | 1,25(OH)2 Vitamin D3
Number analyzed (Participants) | 104 | 100
mmol/L | 1.27 (0.39) | 1.25 (0.33)
Statistical Analysis 1: Comparison: Vitamin D2; The levels of blood phosphorus were compared between the 24th month of following up and the baseline in group Vitamin D2; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1,25(OH)2 Vitamin D3; The levels of blood phosphorus were compared between the 24th month of following up and the baseline in group 1,25(OH)2 Vitamin D3, respectively; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Vitamin D2 vs 1,25(OH)2 Vitamin D3; The levels of blood phosphorus at the 24th month of following up were compared between two groups; Test type: Superiority or Other; p = 0.694, t-test, 2 sided — t=0.394

5. Primary Outcome: The Blood Levels of Intact Parathyroid Hormone at the 24th Month of Following up.
Description: The blood levels of intact parathyroid hormone (iPTH) at the 24th month of following up will be detected.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vitamin D2 | 1,25(OH)2 Vitamin D3
Number analyzed (Participants) | 104 | 100
pg/ml | 96.5 (87.1) | 108.1 (134.0)
Statistical Analysis 1: Comparison: Vitamin D2; The levels of blood iPTH were compared between the 24th month and the baseline in group Vitamin D2; Test type: Superiority or Other; p = 0.179, t-test, 2 sided
Statistical Analysis 2: Comparison: 1,25(OH)2 Vitamin D3; The levels of blood iPTH were compared between the 24th month and the baseline group 1,25(OH)2 Vitamin D3, respectively; Test type: Superiority or Other; p = 0.106, t-test, 2 sided
Statistical Analysis 3: Comparison: Vitamin D2 vs 1,25(OH)2 Vitamin D3; The levels of blood iPTH at the 24th month of following up were compared between two groups; Test type: Superiority or Other; p = 0.463, t-test, 2 sided — t=-0.736

ADVERSE EVENTS:
Arm/Group | Vitamin D2 | 1,25(OH)2 Vitamin D3
Serious Adverse Events (participants affected / at risk) | 13/104 | 10/100
Other Adverse Events (participants affected / at risk) | 10/104 | 8/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D2 (N=104) | 1,25(OH)2 Vitamin D3 (N=100)
AMI (Cardiac disorders) | 2 | 3
congestive heart failure (Cardiac disorders) | 1 | 3
Stroke (Nervous system disorders) | 3 | 2
In patient (General disorders) | 7 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D2 (N=104) | 1,25(OH)2 Vitamin D3 (N=100)
Renal replacement therapy (Renal and urinary disorders) | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No